CLINICAL TRIAL: NCT01582841
Title: Integrating Genetic Testing for Lynch Syndrome in a Managed Care Setting
Acronym: HNPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Case Western Reserve University (Other); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R01CA140377-01A2 (NIH)
Record Dates: First submitted 2011-12-15; First posted 2012-04-23 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer; Lynch Syndrome
Keywords: Colon Cancer; Lynch Syndrome; Genetic Screening
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSI testing (Experimental): All individuals in the intervention arm who consent to participate in the HNPCC screening will have their tumors evaluated for MSI following surgery. Those with MSI-H results will receive a genetic counseling informational call.
  Interventions: Procedure: MSI screening test
- Usual care (No Intervention): These patients will be treated as usual by their oncologist and medical team. These patients receive a follow up letter a year after randomization, alerting them to the availability of clinical Lynch Syndrome screening.

INTERVENTIONS:
Procedure: MSI screening test — All individuals in the intervention arm who consent to participate in the HNPCC screening will have their tumors evaluated for MSI.
  Arms: MSI testing

SUMMARY:
The investigators research mobilizes the resources of an integrated health-delivery system with extensive electronic clinical data to implement and evaluate a new strategy to maximize screening of Colorectal Cancer (CRC) patients for Lynch Syndrome.

DETAILED DESCRIPTION:
Screening tests for Hereditary Non-Polyposis Colorectal Cancer (HNPCC) [also called Lynch Syndrome], are among the few available validated genetic tests that have been recommended as an evidence-based practice that can save lives. However, more than half of patients who meet well-established and accepted screening criteria do not receive screening. This is a critical failure for patients and for the health-care delivery system because HNPCC mutation carriers are at exceptionally high risk for colorectal and other HNPCC-related cancers, and because clinical strategies can prevent future cancers, or provide early detection, for individuals affected with HNPCC and their relatives. HNPCC testing is also cost-effective compared to treating individuals with a diagnosis of colorectal cancer (CRC).

To address this shortfall in practice, our proposed research mobilizes the resources of an integrated health-delivery system with extensive electronic clinical data to implement and evaluate a new strategy to maximize screening of CRC patients for HPNCC. The Evaluation of Genomic Applications in Practice and Prevention (EGAPP) working group recommended that all newly diagnosed CRC patients be screened for HPNCC, but was not able to recommend a best-strategy to accomplish this aim. Therefore, using the Practical Robust Implementation and Sustainability Model (PRISM), developed by one of our co-investigators, to guide the analyses, the investigators will:

Aim #1: Conduct a randomized controlled trial to determine the effectiveness of a universal laboratory test-based HNPCC screening program compared to the current practice of physician referral and self-referral.

Aim #2: Elucidate patient, provider, and system factors important to success of implementation.

Aim #3: (revised and approved during year 1): To create, refine, and disseminate an implementation guide for HNPCC screening by combining the results from Aims 1-2 and the perspectives from informant interviews of key staff at future diverse dissemination-implementation sites: Case Western Reserve University, Oregon Health & Sciences University, MD Anderson Cancer Center, Dana-Farber Cancer Institute, Kaiser Permanente Georgia, Kaiser Permanente Hawaii, and Safety Net West Clinics. Addition to Aim 3: We will contribute materials to the LSSN website for dissemination of implementation materials.

This study aims to evaluate implementation of a novel HNPCC screening program and assess, for all stakeholders, facilitators and barriers to program implementation and success. Results from this study will help achieve the Healthy People 2020 objective of reducing CRC mortality. It will add to the growing literature in the increasingly important area of translating research findings into real-world practice, a subject of the NIH Roadmap. Many of the findings will be useful in other clinical areas and will be broadly applicable to other health care organizations aiming to improve access to genetic tests for cancers.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Kaiser Permanente member
3. Referral or scheduled colon surgery
4. No known cognitive impairments (e.g., Alzheimer's Disease) that would impact the ability to be consented
5. English speaker
6. Diagnosis of colon cancer

Exclusion Criteria:

1. Under the age of 18
2. Known cognitive impairment
3. Inability to speak/understand English
4. On the research exclusion list
5. Known Lynch syndrome
6. No diagnosis of colon cancer
7. In hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Implementation effectiveness | All patients will be followed up to 5 years. Most active participation and chart review will take place within one year of surgery.
  The primary outcomes to assess implementation effectiveness are: number of patients who receive HNPCC screening test results; number of physicians who receive their patients HPNCC screening test results; completion of the educational session at three months of follow-up; and number of patients with MSI-H (microsatellite instability-high) test results who are contacted by medical genetics.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina AB Goddard, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States